CLINICAL TRIAL: NCT03855527
Title: Effectiveness of Silver Diamine Fluoride as Cavity Disinfectant After Atraumatic Restorative Treatment in Primary Teeth: A Randomized Clinical Trial
Brief Title: Effectiveness of Silver Diamine Fluoride as Cavity Disinfectant After Atraumatic Restorative Treatment in Primary Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Clinical Instructor and statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDF as cavity disinfectant
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Dental Caries
Keywords: Atraumatic Restorative Treatment; Chlorhexidine; Silver Diamine Fluoride; Primary Teeth
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride; Chlorhexidine; Disinfection

STUDY DESIGN:
Intervention Model Description: This study is a three arm randomized controlled clinical trial, where children indicated for Atraumatic Restorative Treatment (ART) will be selected.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The operator will not be blinded to the type of treatment as each antibacterial agent has different consistency, color and application technique. However the expert assessing the microbiologic sample and statistician will be blinded to the treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silver Diamine Fluoride (SDF) group (Experimental): Atraumatic restorative technique will be performed. Then the cavities will be dried with a gentle flow of compressed air. One drop of silver diamine fluoride (Advantage Arrest Silver Diamine Fluoride 38% - Bottle) will be dispensed into a dappen dish. A micro brush will be bent, dipped into SDF and dabbed on the side of the dappen dish to remove excess liquid before application. SDF will be applied directly to affected tooth surface and dried with gentle flow of compressed air for 1 minute. Excess SDF will be removed with cotton roll. Teeth will be restored with glass ionomer cement (GC Fuji IX).
  Interventions: Drug: Silver Diamine Fluoride
- Chlorhexidine group (Active Comparator): Atraumatic restorative treatment will be performed. Then, the cavities will be disinfected by placing a cotton pellet soaked in chlorhexidine solution (Consepsis®2% Chlorhexidine Antibacterial Solution) for 1 minute, air dried and restored using glass ionomer cement.
  Interventions: Drug: Chlorhexidine
- Atraumatic Restorative Treatment without Disinfection (Sham Comparator): Cavities will be cleaned according to the ART approach.The cavity will be enlarged if needed using sterile hatchet.The carious dentin will be removed with excavators starting at the enamel-dentine junction. The unsupported thin enamel will be fractured off with the hatchet. The caries will be removed carefully until firm dentin is reached (physically resistant to hand excavation). The cavity will be cleaned with wet cotton pellets. Cavities will be restored immediately using conventional glass ionomer cement. All the cavities in the 3 groups will be temporary restored with glass ionomer cement handled according to manufacturer's instructions, however acid etching will not be carried out in order to make sample collection easier following the experimental period.
  Interventions: Procedure: Atraumatic Restorative Treatment without Disinfection

INTERVENTIONS:
Drug: Silver Diamine Fluoride — SDF will be applied as a cavity disinfected after atraumatic restorative technique (Antimicrobial effect)
  Other Names: SDF
  Arms: Silver Diamine Fluoride (SDF) group
Drug: Chlorhexidine — Chlorhexidine will be applied as a cavity disinfected after atraumatic restorative technique (Antimicrobial effect)
  Other Names: CHG
  Arms: Chlorhexidine group
Procedure: Atraumatic Restorative Treatment without Disinfection — Atraumatic Restorative Technique will be performed without cavity disinfection
  Arms: Atraumatic Restorative Treatment without Disinfection

SUMMARY:
The purpose of this study is to evaluate the effectiveness of silver diamine fluoride (SDF) compared to chlorhexidine (CHX) as a cavity disinfectant in primary molars after Atraumatic Restorative Treatment approach (ART).

DETAILED DESCRIPTION:
This study is a three arm randomized controlled clinical trial, where children with an age range of 4-6 years indicated for Atraumatic Restorative Treatment (ART) are selected from the outpatient clinic of Pediatric Dentistry and Public Health Department, Faculty of Dentistry, Alexandria University after securing necessary consents. Sixty teeth are randomly allocated into 3 groups of Atraumatic restorative treatment approaches. Group I is assigned to silver diamine fluoride as an antibacterial agent, Group II is assigned to chlorhexidine as an antibacterial agent, and Group III serves as a negative control.

ELIGIBILITY:
Inclusion Criteria:

* Children free of any systemic disease or special health care needs.
* Class I cavity involving dentin in primary molars.
* Lesion wide enough to allow access of instruments.
* Informed consent fulfilled.

Exclusion Criteria:

* Signs of irreversible pulpitis or pulp necrosis.
* Patients allergic to silver products.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Microbiological assessment of total viable bacterial count | First day (baseline)
  The first dentin sample will be collected with a sterile spoon excavator from the firm dentin in the center of the cavity. Two microliters of the samples collected will be inoculated on blood agar for total viable count.
Microbiological assessment of streptococcus mutans count | First day (baseline)
  The first dentin sample will be collected with a sterile spoon excavator from the firm dentin in the center of the cavity. Two µl of the samples will be inoculated on mitis salivarius agar supplemented with 15 percent sucrose and bacitracin (0.2 U/ml) for selective isolation of Streptococcus mutans.
Microbiological assessment of lactobacilli count | First day (baseline)
  The first dentin sample will be collected with a sterile spoon excavator from the firm dentin in the center of the cavity.Two µl of the samples will be inoculated on Rogosa agar, a medium selective for Lactobacilli.
Change in the total viable count. | 14 days
  A second dentin sample will be taken from the same position with a sterile round bur for bacteriologic assessment.
Change in the lactobacilli count. | 14 days
  A second dentin sample will be taken from the same position with a sterile round bur for bacteriologic assessment.
Change in the streptococcus mutans count. | 14 days
  A second dentin sample will be taken from the same position with a sterile round bur for bacteriologic assessment.

SECONDARY OUTCOMES:
Clinical changes in the dentin color | 14 days
  Restoration will be removed and the dentin will be checked using visual-tactile method of examination.
Clinical changes in the dentin consistency | 14 days
  Restoration will be removed and the dentin will be checked using visual-tactile method of examination.

CONTACTS AND LOCATIONS:
Overall Officials: Lina A Matar, BDS, Principal Investigator — Alexandria University; Karin ML Dowidar, PhD, Study Director — Alexandria University; Dalia AM Talaat, PhD, Study Director — Alexandria University; Dina AE Kholeif, PhD, Study Director — Faculty of Medicine, Alexandria Univerity
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Joshi JS, Roshan NM, Sakeenabi B, Poornima P, Nagaveni NB, Subbareddy VV. Inhibition of Residual Cariogenic Bacteria in Atraumatic Restorative Treatment by Chlorhexidine: Disinfection or Incorporation. Pediatr Dent. 2017 Jul 15;39(4):308-312. PMID 29122072
- [Background] Horst JA, Ellenikiotis H, Milgrom PL. UCSF Protocol for Caries Arrest Using Silver Diamine Fluoride: Rationale, Indications and Consent. J Calif Dent Assoc. 2016 Jan;44(1):16-28. PMID 26897901
- [Background] Innes NP, Frencken JE, Bjorndal L, Maltz M, Manton DJ, Ricketts D, Van Landuyt K, Banerjee A, Campus G, Domejean S, Fontana M, Leal S, Lo E, Machiulskiene V, Schulte A, Splieth C, Zandona A, Schwendicke F. Managing Carious Lesions: Consensus Recommendations on Terminology. Adv Dent Res. 2016 May;28(2):49-57. doi: 10.1177/0022034516639276. PMID 27099357
- [Background] Massara ML, Alves JB, Brandao PR. Atraumatic restorative treatment: clinical, ultrastructural and chemical analysis. Caries Res. 2002 Nov-Dec;36(6):430-6. doi: 10.1159/000066534. PMID 12459616
- [Background] Bjorndal L, Larsen T, Thylstrup A. A clinical and microbiological study of deep carious lesions during stepwise excavation using long treatment intervals. Caries Res. 1997;31(6):411-7. doi: 10.1159/000262431. PMID 9353579
- See also: Manual for the atraumatic restorative treatment approach to control dental caries. — http://vida.gt/clinica/doctores/wp-content/uploads/sites/2/2014/07/ART_Manual_English.pdf
- See also: Use of Silver Diamine Fluoride for Dental Caries Management in Children and Adolescents, Including Those with Special Health Care Needs. reference manual of American academy of pediatric dentistry — http://www.aapd.org/media/policies_guidelines/g_sdf.pdf